CLINICAL TRIAL: NCT06568731
Title: A PHASE 1, OPEN- LABEL STUDY TO EVALUATE THE MULTIPLE DOSE PHARMACOKINETICS OF DANUGLIPRON FOLLOWING ORAL ADMINISTRATION IN OTHERWISE HEALTHY ADULT PARTICIPANTS WITH OVERWEIGHT OR OBESITY
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Danuglipron Are Taken up Into the Blood in Otherwise Healthy Adults With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3421069; NCT06568731 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Overweight; Obesity; Danuglipron; GLP-1; Overtly healthy
MeSH Terms: conditions — Obesity; Overweight | interventions — danuglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participants will receive multiple doses of danuglipron
  Interventions: Drug: Danuglipron

INTERVENTIONS:
Drug: Danuglipron — Danuglipron oral tablets
  Other Names: PF-06882961

SUMMARY:
The purpose of this study is to learn the following about the study medicine, danuglipron, after multiple days of dosing in healthy adults who are overweight or obese:

* how the study medicine, danuglipron, is taken up into the blood
* about the safety and tolerability of danuglipron

The total number of weeks of the study is about 15 (about 4 months).

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years of age or older
* Body mass index (BMI) of ≥25.0-45.4 kg/m2; and a total body weight >50 kg (110 lb)

Key Exclusion Criteria:

* Evidence or history of any clinically significant medical conditions or laboratory abnormality
* Any condition possibly affecting drug absorption
* Known intolerance/hypersensitivity to a GLP-1R agonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-08-23 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Steady-state area under the concentration-time profile from time zero to 24 hours (AUC24) for danuglipron | Predose to 24 hours post danuglipron administration
Steady-state maximum observed concentration (Cmax) for danuglipron | Predose to 24 hours post danuglipron administration
Steady-state time to reach maximum observed concentration (Tmax) for danuglipron | Predose to 24 hours post danuglipron administration

SECONDARY OUTCOMES:
Number of participants reporting Treatment Emergent Adverse Events (TEAEs) | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant clinical laboratory abnormalities | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant vital sign abnormalities | From baseline up to 28-35 days post last dose taken
Change from baseline in body weight | From baseline up to 28-35 days post last dose taken
Number of participants reporting clinically significant changes ECG abnormalities | From baseline up to 28-35 days post last dose taken

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421069